CLINICAL TRIAL: NCT02890719
Title: Pilot Study Evaluate Efficacy of Grazoprevir + Elbasvir for 12 or 16 Weeks in Liver Transplant Recipients.
Acronym: EGRADICATE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Impossibility of supplying the medication in research of the study by the pharmaceutical company that gave it to the trial
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Xavier Forns, Fundacion Clinic per a la Recerca Biomédica
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGRADICATE; 2015-005453-13 (EudraCT Number)
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Liver Transplantation; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotype 1B (Experimental): treatment 12 weeks
  Interventions: Drug: Grazoprevir 100 mg/day; Drug: Elbasvir 50 mg/d
- Genotype 1A and 4 (Experimental): treatment 16 weeks
  Interventions: Drug: Grazoprevir 100 mg/day; Drug: Elbasvir 50 mg/day; Drug: Ribavirin 1200 mg/day

INTERVENTIONS:
Drug: Grazoprevir 100 mg/day — Grazoprevir 100 mg/ day 12 weeks
  Other Names: J05AX68 100 mg
  Arms: Genotype 1B
Drug: Elbasvir 50 mg/d — Elbasvir 50 mg/day 12 weeks
  Other Names: J05AX68 50mg
  Arms: Genotype 1B
Drug: Grazoprevir 100 mg/day — Grazoprevir 100 mg/day 16 weeks
  Other Names: J05AX68 100 mg
  Arms: Genotype 1A and 4
Drug: Elbasvir 50 mg/day — Elbasvir 50 mg/d 16 weeks
  Other Names: 50mg J05AX68
  Arms: Genotype 1A and 4
Drug: Ribavirin 1200 mg/day — Ribavirin 1200 mg/day 16 weeks
  Other Names: J05AB04 1200 mg/d
  Arms: Genotype 1A and 4

SUMMARY:
Pilot, single center, open-label study to evaluate the efficacy and tolerability of Grazoprevir and Elbasvir in HCV GT1 and 4 liver transplant recipients.30 liver transplant recipients with hepatitis C recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 78 year-old.
* Previous liver transplantation(more than 6 month).
* Genotype 1 and 4 infection.
* Hepatitis C recurrence defined by the presence of abnormal liver function test, positive HCV-RNA, histological signs of hepatitis C recurrence.
* Viral load ≥10000UI/mL.
* Immunosuppression with tacrolimus and/or mycophenolate (Prednisone use is allowed at low dose, ≤10 mg/d).
* Treatment naïve or treatment experienced (Peg-RBV or triple therapy).

Exclusion Criteria:

* Genotype 2, 3, 5 or 6 infection.
* Decompensated cirrhosis defined by the presence of actual or previous history of clinical decompensation including ascites, hepatic encephalopathy, variceal bleeding or spontaneous bacterial peritonitis, or a Child-Pugh B or C.
* Hepatocellular carcinoma after liver transplantation.
* Total bilirubin > 3 mg/dL.
* Immunosuppression with cyclosporine or an mTOR inhibitor (everolimus or sirolimus).
* Severe extrahepatic diseases: cardiovascular, respiratory, cerebrovascular and poorly controlled diabetes.
* Platelets < 75 x 109 cells/L.
* Neutrophil count < 0.5 x 109 cells/L.
* Hemoglobin < 9 g/dL.
* Albumin < 3g/dL.
* HIV infection.
* Hepatitis B infection.
* Active intake of toxic amounts of alcohol or recreational drugs.
* Females who are pregnant, become to be pregnant or breastfeeding or males whose partners are pregnant, become to be pregnant or breastfeeding.
* Intake of disallowed medications including(but not limited to):

  1. Antibiotics: clarithromycin, erythromycin, telithromycin, nafcillin, rifampin
  2. Antifungals: itraconazole, ketoconazole, voriconazole
  3. Antihypertensives: nifedipine
  4. Anticonvulsants: carbamazepine, phenytoin, phenobarbital
  5. Bosentan
  6. Modafinil
  7. St.Jonh's Wort
  8. Immunosuppressants: cyclosporin, everolimus, sirolimus
  9. Diabetes agents: glibenclamide, glyburide
  10. Lipid lowering agents: gemfibrozil
  11. Eltrombopag
  12. Lapatinib
  13. HIV medications: efavirenz, etravirine, all ritonavir boosted and unboosted HIV protease inhibitors
  14. Statins: simvastatin, fluvastatin, rosuvastatin at doses greater than 10 mg/d, atorvastatin at doses greater than 10 mg/d.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 12 weeks post-treatment
  Sustained virological response 12 w (SVR24) defined as HCV-RNA undetectable at post-treatment week 12.

SECONDARY OUTCOMES:
Sustained virological response | 4 weeks and 24 weeks post-treatment
  Sustained virological response 12 ( SVR12) defined as HCV-RNA undetectable at post-treatment weeks 4 and , 24 respectively.
To evaluate the beneficial effects of antiviral therapy on renal function. | 24 weeks post-treatment
  creatinine sample analyses blood analyses in all visits
To assess the impact of therapy in kidney function. | 24 weeks post-treatment
  Elevation Transaminases blood analyses in all visits
Tolerability of this combination in liver transplant recipients. | Every visit
  Serious advers events evaluation

IPD SHARING:
Plan to Share IPD: No